CLINICAL TRIAL: NCT02288507
Title: Phase I Study of Sorafenib Concurrent With Yttrium-90 Transarterial Radioembolization in Patients With Advanced Hepatocellular Cancer
Brief Title: Sorafenib Concurrent With Yttrium-90 Transarterial Radioembolization in Patients With Advanced Hepatocellular Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed due to no accrual
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Jared Acoba, Principal Investigator, University of Hawaii
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acoba 2014 -1
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Cancer
Keywords: sorafenib, yttrium-90 radioembolization
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib & Yttrium-90 radioembolization (Experimental): Sorafenib dose de-escalation starting at 400mg PO BID starting on Day1 Yttrium-90 radioemoblization on Day 14
  Interventions: Drug: Sorafenib; Radiation: yttrium-90 radioembolization

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400mg PO BID for Cohort 1, if 2 or more patients with dose-limiting toxicity toxicity (DLT), Chort -1 is sorafenib 200mg PO BID, if 2 or more patients with DLT, sorafenib 200mg PO daily
  Other Names: Nexavar; Bay 43-9006 tosylate; Bay 54-9085
Radiation: yttrium-90 radioembolization — Yttrium-90 SIR-Spheres microspheres are instilled through a catheter into a branch of the hepatic artery
  Other Names: SIR-Spheres microspheres

SUMMARY:
This study evaluates the safety and efficacy of administering sorafenib concurrent with yttrium-90 radioembolization to patients with advanced hepatocellular cancer.

DETAILED DESCRIPTION:
Studies in Asia of unresectable hepatocellular cancer (HCC) demonstrated that sorafenib could be administered safely at 400mg twice a day (BID) when initiated 14 days following radioembolization (RE). However, the ideal sequence of RE and sorafenib may not be completely elucidated, the two treatments given concurrently may be more effective than the sequential approach studied in the Asian trials. Preclinical models have demonstrated that sorafenib acts synergistically with radiation, increasing apoptosis. Furthermore, case reports suggest profound responses in patients who have received sorafenib concurrent with transarterial radioembolizatoin (TARE) as evidenced by improvement in symptoms, >80% decrease in alpha fetoprotein (AFP), and conversion from unresectable to resectable. Sorafenib concurrent with TARE may take advantage of the synergistic relationship between the two therapies and prove to be a more effective treatment strategy than sequential administration of TARE and sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HCC or clinical diagnosis by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic subjects is required. m)
* Barcelona Clinic Liver Cancer Stage B or C. Segmental and subsegmental portal vein thrombosis is allowed.
* Metastatic disease is allowed if investigator feels liver directed therapy could offer palliative benefit (i.e., minimal extrahepatic tumor burden)
* No evidence of cirrhosis or cirrhosis grade of Child-Pugh class A or B7. Eligibility
* Have at least one tumor lesion that can be accurately measured according to Response Evaluation Criteria in Solid Tumor (RECIST v1.1).
* Consultation with interventional radiologist and deemed an appropriate candidate for TARE.
* Prior local therapy, such as surgery, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation is allowed if the index lesion(s) remains outside of the treatment field or has progressed since prior treatment. Local therapy must have been completed at least 4 weeks prior to the baseline scan.
* Prior yittrium-90 transarterial radioembolization (TARE) or sorafenib not allowed
* Patient must be informed of the investigational nature of this study, sign and give written informed consent in accordance with institutional and federal guidelines.
* Age ≥ 18 years.
* Eastern Cooperative Group (ECOG) performance status ≤ 1.
* Have adequate hematologic function as documented by an absolute neutrophil count (ANC) ≥ 1000/ul, platelet count ≥ 60,000/ul, and hemoglobin ≥ 8.5 mg/dl obtained within 28 days prior to registration.
* Have adequate hepatic function, as determined by the following tests measured within 28 days prior to registration: serum bilirubin ≤ 2 x upper limit of normal (ULN); serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) ≤ 5 x the institutional upper limit of normal (IULN).
* Have adequate renal function, as determined by the following tests measured within 28 days prior to registration: serum creatinine ≤ 1.5 x ULN OR a measured creatinine clearance or calculated creatinine clearance ≥ 50 mL/min.
* Have a life expectancy of ≥12 weeks
* Must be able to swallow oral medications.
* Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.

Exclusion Criteria:

* Known or suspected allergy or hypersensitivity to sorafenib.
* Any malabsorption condition.
* Must not have known brain metastases.
* No concurrent anticancer chemotherapy or local therapy.
* No concurrent herbal or unconventional therapy (e.g., St. John's Wort)
* Pregnant or nursing women
* No prior radiation therapy to the liver
* Inability to perform y90 TARE due to: (1) inability to catheterize the hepatic artery, (2) portal vein thrombosis/occlusion without the ability to perform selective infusion, (3) Tecnetium-99m macro-aggregated albumin hepatic artery perfusion scintigraphy shows unfavorable shunt fraction between the liver and the pulmonary parenchyma as determined by the interventional radiologist, or (4) other contraindication to TARE identified by interventional radiologist.
* Women/men of reproductive potential unwilling or unable to use an effective contraceptive method
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 3 years.
* History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within 6 months.
* Concurrent severe or uncontrolled medical disease (i.e., active systemic infection, diabetes, coronary artery disease, congestive heart failure) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of concurrent sorafenib and yttrium-90 transarterial radioembolization (TARE) for patients with advanced hepatocellular cancer as measures by Adverse events | 2 months
  All patients will be monitored and evaluated for clinical toxicities during the treatment period and queried at each follow-up visit for Adverse Events (AEs). Patients may volunteer information concerning AEs. All AEs will be graded by using the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).

SECONDARY OUTCOMES:
Efficacy of concurrent sorafenib and yttrium-90 transarterial radioembolization (TARE) for patients with advanced hepatocellular cancer as measured by response rate, time to progression (TTP), progression free survival (PFS), overall survival (OS) | 1 year
  Response: Response will be evaluated by contrast enhanced MRI or CT and response rates will be reported separately as measured by RECIST and mRECIST criteria. Duration of response will also be measured according to RECIST and mRECIST guidelines.
  Survival: The time to progression, progression free survival, and overall survival will be measured. TTP and PFS will be calculated based on progression as defined by RECIST and mRECIST and both intervals will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Acoba, MD, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No